CLINICAL TRIAL: NCT04491448
Title: Acceptability of Social Risk Screening in Adult Primary Care
Brief Title: Acceptability of Social Risk Screening
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Steven M. Albert, Professor, University of Pittsburgh
Other Study IDs: STUDY20010212
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Primary Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Social needs screening — Interview and referral for non-medical health-related social needs

SUMMARY:
Social risk screening asks patients to provide information on health-related social needs that are non-medical but affect health. These include housing stability, food security, reliable medical transportation, consistent utilities service (heat, light, water), and interpersonal safety. This research will determine the acceptability of such screening in adult patients who attend a primary care clinic in-person or via a telemedicine visit, the level of social need in patients, and how to flag such information for care, planning, and follow up.

DETAILED DESCRIPTION:
This study will evaluate the acceptability of social risk screening among adult patients seen in the General Internal Medicine Offices (GIMO) at Montefiore Hospital. The research will enroll patients using the resident clinic, which provides medical care to lower-income patients as well as other patients. The study will be limited to new patients or patients receiving routine follow-up care.

Acceptability will be assessed by (i) the proportion of patients completing the screen among those approached; (ii) the proportion of screening questions completed; and (iii) the proportion of patients willing to complete the screening over the phone (a) by interviewer or (b) on via website using Qualtrics.

The representativeness of the sample will be assessed by comparing the participant sample to aggregate clinic demographic characteristics and deidentified Epic EHR indicators using an honest broker.

The survey instrument is the CMS Accountable Care Communities instrument. It includes patient indicators (demography) and appraisals of care (e.g., trust) that will allow assessment of correlates of social need and acceptability of screening in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18+
2. New patient or routine physical exam, GIMO clinic, Montefiore Hospital

Exclusion Criteria:

1. Unable to provide verbal informed consent
2. Unable to complete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for a routine physicals or new patient visits
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of social needs screening in medical encounter | One-time interview, 20-25 minutes
  Proportion reporting social needs relevant to medical care

SECONDARY OUTCOMES:
Effects of reported social needs on medical utilization and patient behavior | One-time interview, 20-25 minutes
  Reports of missed appointments and need for social work referrals

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Albert, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available to other researchers and students who approach the investigators and prepare detailed analytic plans. The Office of Sponsored Programs will review requests to share de-identified research data/materials to determine whether an agreement needs to be executed.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 Months after study completion
Access Criteria: Contact PI